CLINICAL TRIAL: NCT03874884
Title: 177Lu-PSMA-617 Therapy and Olaparib in Patients With Metastatic Castration Resistant Prostate Cancer
Acronym: LuPARP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Peter Mac project no.18/216
Record Dates: First submitted 2019-02-28; First posted 2019-03-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-PSMA + olaparib (Experimental): Patients will receive a fixed 7.4 GBq of 177Lu-PSMA every 6 weeks together with olaparib on days 2-15 of each cycle. A cycle is 42 days long. Patients will receive 6 cycles of treatment.
  Interventions: Drug: Olaparib; Combination Product: 177Lu-PSMA

INTERVENTIONS:
Drug: Olaparib — During dose escalation doses of olaparib that can be administered are 50mg BD D2-15, 100mg BD D2-15, 150mg BD D2-15, 200mg BD D2-15,250mg BD D2-15, 300mg BD D2-15, 200mg BD D4-14, 300mg BD D-4-14 or 400mg D-4-18 of a 42 day cycle for up to 6 cycles.
  The recommended phase 2 dose of olaparib will be used in 2 consecutive dose expansion cohorts. The first cohort will received the recommended phase 2 dose of Olaparib on D4-14 of a 42 day cycle. Patients enrolled in the second dose expansion cohort will receive Olaparib continuously from cycle 1 day -4 to cycle 6 day 42.
Combination Product: 177Lu-PSMA — A fixed 7.4Gbq administered activity of 177Lu-PSMA will be given 6 weekly for up to 6 cycles.

SUMMARY:
This phase 1 dose-escalation and dose-expansion study is designed to evaluate the safety and tolerability of olaparib in combination with 177Lutetium-Prostate Specific Membrane Antigen (177 Lu-PSMA) in patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This phase 1, open label, multicentre, dose-escalation and dose-expansion study is designed to evaluate the safety and tolerability of olaparib in combination with 177Lu-PSMA in patients with mCRPC. Patients with mCRPC who have previously progressed on a novel AR targeted agent (abiraterone and/or enzalutamide and/or apalutamide) and have not had prior exposure to platinums, PARP inhibitors or 177Lu-PSMA will be eligible for the study. Patients can have had prior exposure to docetaxel in the chemotherapy naïve setting or castrate setting.

Patients will be enrolled in two stages: a dose escalation and a dose expansion phase. The clinical and translational outcomes from this study will inform the design of future phase 2/3 clinical trials of this combination.

This is a single arm study where patients will receive 177Lu-PSMA and olaparib for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria for study entry:

1. Patient must be ≥ 18 years of age and must have provided written informed consent.
2. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell differentiation.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (see Appendix 1).
4. For dose escalation (dose levels 1-9) and expansion cohorts, patients must have had at least one prior line of taxane (docetaxel) chemotherapy either in the hormone sensitive or castrate resistant setting unless the patient is deemed medically unsuitable for chemotherapy. If a patient has had docetaxel chemotherapy twice, this will be considered one line. For the continuous olaparib dose cohort (DE #2) patients can have had docetaxel however this is not required for eligibility.
5. Patients must have progressed on a second generation AR targeted agent (e.g. enzalutamide, abiraterone, darolutamide and/or apalutamide). Determination of disease progression on second generation AR targeted agent will be made by the local investigator.
6. Patients must have progressive disease for study entry. This is defined by PCWG3 as any one of the following:

   * PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement. The PSA value at screening should be ≥ 10ng/ml.
   * Soft tissue or visceral disease progression as per RECIST 1.1 criteria (see Appendix 2)
   * Bone progression: ≥ 2 new lesions on bone scan (Appendix 2)
7. At least 3 weeks since the completion of surgery or radiotherapy prior to registration. Any clinically relevant sequelae from the surgery or radiotherapy must have improved to grade 1 prior to registration.
8. Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist). Patients without prior surgical castration must be currently taking and willing to continue luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) therapy throughout the duration of study treatment.
9. Serum testosterone levels ≤ 50ng/dL (≤ 1.75nmol/L) within 28 days before registration.
10. Imaging evidence of metastatic disease documented with either bone scan or CT scan (Appendix 2).
11. Prior prostate cancer vaccine therapy, radiation therapy, systemic therapies, diethylstilboestrol (DES) or other estrogens, bicalutamide, flutamide or nilutamide are allowed up to 28 days prior to trial registration. Note: bicalutamide, flutamide or nilutamide must be discontinued within 4 weeks of registration.
12. Significant PSMA avidity on 68Ga/18F-PSMA PET/CT, defined as a minimum uptake of SUVmax 15 at a site of disease, and SUVmax > 10 at other sites of disease ≥10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact).
13. Patients must have a life expectancy ≥ 24 weeks.
14. Patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see section 11.7.4 for acceptable methods).
15. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled assessments including completing Patient Reported Outcomes (PRO) instruments.
16. Patients must have adequate bone marrow, hepatic and renal function documented within 28 days prior to registration, defined as:

    * Haemoglobin ≥ 100 g/L independent of transfusions (no red blood cell transfusion in last 8 weeks)
    * Absolute neutrophil count ≥ 1.5x109/L
    * Platelets ≥ 150 x109/L
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome where this applies for the unconjugated bilirubin.
    * Aspartate transaminase (AST) (SGOT) and alanine transaminase (ALT) (SGPT) ≤ 2.5 x ULN if there is no evidence of liver metastasis or ≤ 5 x ULN in the presence of liver metastases.
    * Albumin ≥ 30 g/L
    * Adequate renal function: patients must have creatinine clearance estimated of ≥ 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test to appendix 5).
17. Patients who are deemed by PSMA imaging to have readily accessible disease will be required to consent to 3 serial tumour biopsies - at screening, post combination treatment (at any time between weeks 2-4) and in the event of disease progression.

Exclusion Criteria:

Patients must not meet any of the following criteria for study entry:

1. Site(s) of disease that are FDG positive with low PSMA expression defined by PSMA SUVmax < 10.
2. Extensive marrow disease defined by a "Super Scan" on bone scintigraphy or diffuse marrow infiltration on PSMA PET.
3. Previous history or presence of brain metastases or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required if there is no clinical history of this.
4. Surgery or radiotherapy within < 3 weeks of registration (except for palliative reasons). Patients must have recovered from any effects of any major surgery.
5. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable for ≥ 4 weeks.
6. Any prior exposure to 177Lu-PSMA, cabazitaxel, platinums, PARP inhibitors, mitoxantrone or cyclophosphamide.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent thromboembolic events (<6 months ago), uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or psychiatric illness/social situations that is likely to impede participation and /or compliance in the study.
8. Persistent toxicities [Common Terminology Criteria for Adverse Event (CTCAE) ≥ grade 2] caused by previous cancer therapy, excluding alopecia.
9. Other malignancies within the previous 2-years other than basal cell or squamous cell carcinomas of skin or other cancers that are unlikely to recur within 24 months.
10. Previous history of interstitial lung disease or non-infectious pneumonitis.
11. Patients with a history or clinical features suggestive of myelodysplastic syndrome / acute myeloid leukaemia.
12. Patients unable to swallow orally administered medications or with gastrointestinal disorders likely to interfere with the absorption of the study medication.
13. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
14. Known hypersensitivity to olaparib or any of the excipients of olaparib.
15. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV1/2). Only need to check this if there is a clinical history. HIV-infected (HIV1/2 antibody-positive) patients may participate if they meet all the following eligibility requirements:

    * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within the past 12 weeks.
    * They must have a CD4 count ≥ 250 cells/µL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/µl over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy-induced bone marrow suppression.
    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/µl during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy.
    * They must have an undetectable viral load and a CD4 count ≥ 250 cells/µL within 7 days of enrolment.
    * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months.
16. Patients with known active hepatitis (i.e. Hepatitis B or C). Only need to check this if there is a clinical history.

    * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
18. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and enzalutamide and 3 weeks for other agents.
19. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
20. Participation in another clinical study with an investigational product or another systemic therapy administered in the last 3 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with mCRPC who are minimally symptomatic and have progressed on at least one line of novel AR targeted agents (e.g. enzalutamide, abiraterone acetate, apalutamide, etc) will be eligible for the study.Patients may have received docetaxel chemotherapy in the treatment naïve or castrate resistant setting. Prior prostate cancer vaccine therapy, radiation therapy, systemic therapies, diethylstilboestrol (DES) or other oestrogens, bicalutamide, flutamide or nilutamide are allowed up to 28 days prior to trial registration (bicalutamide, flutamide or nilutamide must be discontinued within 4 weeks of registration). Patients already receiving anti-bone resorptive therapy for management of skeletal related events (SREs) are permitted to continue with this treatment.
Enrollment: 70 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting toxicities (DLTs) | Dose escalation phase is expected to be completed 11 months from the time the first patient is recruited.
  A DLT is defined as a toxicity that prevents further administration of the trial treatment at that dose level.
  Each cohort of 3 patients be assessed for DLTs in the first 6 weeks (cycle 1) of treatment and a dose for the next cohort will be determined.
Maximum Tolerated dose (MTD) | Dose escalation phase is expected to be completed 11 months from the time the first patient is recruited.
  The MTD is defined as the highest dose level at which the incidence of DLT was less than 2/6.
Recommended Phase 2 Dose (RP2D) | Upto 30 months from the time the first patient is recruited.
  After the MTD is established, additional patients will be treated at the MTD. Safety and efficacy data from the study will be used to define the RP2D.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. | Through study completion, up until 18 months after the last patient commences treatment.
  Safety of the combination will be measured by AEs and SAEs.
Radiographic progression-free survival (rPFS) | Through study completion, up until 18 months after the last patient commences treatment.
  rPFS is defined as the time from treatment initiation to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first. The radiographic progression will be assessed by the investigator per RECIST1.1 for soft tissue and PCWG3 for bone lesions.
PSA progression free survival (PSA-PFS) | Through study completion, up until 18 months after the last patient commences treatment.
  PSA-PFS is defined as the time from treatment initiation to the date of PSA progression per PCWG3 or death due to any cause, whichever occurs first. The date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2ng/mL or more from the nadir is documented. For patients who have an initial PSA decline during treatment, this must be confirmed by a second value 3 or more weeks later.
Objective response rate (ORR) by RECIST1.1 in patients with measurable disease | Through study completion, up until 18 months after the last patient commences treatment.
  Objective Response (OR) is only applicable for the subset of patients with measurable disease by RECIST1.1. OR is defined as a partial response (PR) or complete response (CR) at any stage from time of commencement of protocol treatment to the time of subsequent systemic anti-cancer treatment. The ORR is calculated as the proportion of patients with a best response of CR or PR.
Overall survival (OS) | Through study completion, up until 18 months after the last patient commences treatment.
  OS is defined as the time from treatment initiation to the date of death due to any cause.
50% PSA response rate (PSA-RR) | Through study completion, up until 78 weeks after the last patient commences treatment.
  PSA will be assessed at baseline and every 6 weeks from cycle 1 day 1 independent of olaparib and 177Lu-PSMA dosing. PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response.
Duration of response (DOR) | Through study completion, up until 18 months after the last patient commences treatment.
  DOR-PCWG3 is defined as the time between the date of first response (CR/PR per RECIST1.1 for soft tissue and PCWG3 for bone lesions) to the date of first documented radiographic progression per RECIST1.1 for soft tissue and PCWG3 for bone lesions or cancer-related death.
Time to treatment response (TTR) in the subset of patients who achieved a 50% PSA response | Through study completion, up until 18 months after the last patient commences treatment.
  TTR-PCWG3 is defined as the time from treatment initiation to the date of the first documented CR or PR per RECIST1.1 for soft tissue and PCWG3 for bone lesions.
Treatment discontinuation due to toxicity | Through study completion, up until 18 months after the last patient commences treatment.
  The number of patients who discontinue treatment at any time due to treatment related toxicity (yes/no for each patient) will be reported.
Rate of treatment discontinuation due to toxicity | Through study completion, up until 18 months after the last patient commences treatment.
  The percentage of patients who discontinue treatment due to treatment related toxicity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Shahneen Sandhu, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No